CLINICAL TRIAL: NCT03074032
Title: Phase I Open-label Single- and Multiple-ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ONC1-0013B in Patients With Progressive Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Safety, Tolerability and Pharmacokinetics of ONC1-0013B in Patients With Progressive Metastatic Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avionco LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-ONC10013B-01
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ONC1-0013B 40 mg (Experimental): ONC1-0013B 40 mg per os daily
  Interventions: Drug: ONC1-0013B
- ONC1-0013B 80 mg (Experimental): ONC1-0013B 80 mg per os daily
  Interventions: Drug: ONC1-0013B
- ONC1-0013B 160 mg (Experimental): ONC1-0013B 160 mg per os daily
  Interventions: Drug: ONC1-0013B
- ONC1-0013B 320 mg (Experimental): ONC1-0013B 320 mg per os daily
  Interventions: Drug: ONC1-0013B

INTERVENTIONS:
Drug: ONC1-0013B — ONC1-0013B per os daily

SUMMARY:
This is a PhaseI, open-label study, Dose-Escalation Study, where tolerated doses will be escalated to the next doses with the safety, tolerability, and PK being evaluated in metastatic castration-resistant prostate cancer (mCRPC) patients. Tumor assessment and PSA values will be evaluated during the study as an additional point.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 years and older.
2. Histologically confirmed diagnosis of prostate cancer
3. Castrate level of testosterone in blood serum < 1,7 nmol/l or < 50 ng/dl
4. PSA level at screening > 2 ng/ml
5. Progression of metastatic CRPC after the chemical castration with gonadotropin-releasing hormone (GnRH) analogue or after the chemical castration and subsequent chemotherapy.
6. The patient's ECOG performance status of 0 - 2
7. Patients previously treated with docetaxel chemotherapy should have received 2 or less prior lines of chemotherapy for mCRPC
8. The expected survival time of not less than 12 weeks

Exclusion Criteria:

1. Prior anticancer therapy:

   * Treatment with chemotherapeutic agents or radiotherapy within 4 weeks prior to screening or preserved toxicities of ≥ II grade according to CTCAE scale, related to prior anticancer therapy (excluding alopecia)
   * Prior antiandrogen therapy: flutamide within 4 weeks prior to screening or bicalutamide within 6 weeks prior to screening
   * Exposure to bisphosphonates is allowed only if the treatment started prior to screening
2. Clinically significant cardiovascular system diseases:
3. Clinically significant central nervous system diseases:
4. History of other significant concomitant diseases which, in the Investigator's opinion, may cause a disease recurrence (i.e. uncontrolled diabetes mellitus)
5. Prior or concomitant therapy:

   * Exposure to drugs which may cause a convulsive state within 4 weeks prior to screening
   * Exposure to treatment with characteristics of CYP3A4 or CYP2D6 inhibitors within 4 weeks prior to screening
   * Exposure to treatment relating to the Class I risk of QT-interval prolongation; exposure to treatment relating to the Class II risk of QT-interval prolongation is allowed if the patient have received not less than 5 half-life periods of flat-dosed treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
DLT within 4 weeks of ONC1-0013B administration (safety and tolerability) | 4 weeks and during the study up to 76 weeks
  Incidence rate and severity of adverse events, changes in laboratory tests

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 28 days
  PK analysis of ONC1-0013B after single and multiple dosage
Area under the plasma concentration versus time curve (AUC) | 28 days
  PK analysis of ONC1-0013B after single and multiple dosage
Elimination half-life (T1/2) | 28 days
  PK analysis of ONC1-0013B after single and multiple dosage
Time-to-peak concentration (tmax) | 28 days
  PK analysis of ONC1-0013B after single and multiple dosage
Steady-State Concentration (Css) | 28 days
  PK analysis of ONC1-0013B after single and multiple dosage
Tumor response | 12 weeks and during the study up to 76 weeks
  RECIST 1.1 criteria and the change of the PSA level

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research Institute of Urology and Interventional Radiology n.a. N.A. Lopatkin (branch of FSBI NMRRC of the Ministry of Health of the Russian Federation), Moscow
  - Medical Radiological Research Center n.a. A.F. Tsyb (branch of FSBI NMRRC of the Ministry of Health of the Russian Federation), Obninsk

IPD SHARING:
Plan to Share IPD: No